CLINICAL TRIAL: NCT05119751
Title: An Investigator-initiated Single Center Randomised Clinical Pilot Study to Compare Tolerability of the Sublingual Versus Vestibular Administration Routes for Birch Pollen, Grass Pollen, Ragweed Pollen, or House Dust Mite Allergy Immunotherapy (AIT)
Brief Title: Vestibular Versus Sublingual Route of AIT Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinique Spécialisée en Allergies de la Capitale (Other)
Collaborators: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT4
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: First month of treatment is taken the vestibular route and the following the sublingual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Birch allergy (Active Comparator): randomised (1:1) to receive vestibular or sublingual birch pollen
  once daily tree 12 SQ-Bet AIT tablet
  Interventions: Drug: tree 12 SQ-Bet
- Grass allergy (Active Comparator): randomised (1:1) to receive vestibular or sublingual grass pollen
  grass 2800 BAU AIT tablet
  Interventions: Drug: GRASS 2800 BAU
- ragweed allergy (Active Comparator): randomised (1:1) to receive vestibular or sublingual ragweed pollen ragweed 12 Amb a 1-U AIT Tablet
  Interventions: Drug: RAGWEED 12 AMB A 1-U
- House dust mite allergy (Active Comparator): randomised (1:1) to receive vestibular or sublingual HDM
  HDM 12 SQ-HDM
  Interventions: Drug: HDM 12 SQ-HDM

INTERVENTIONS:
Drug: tree 12 SQ-Bet — DAILY DOSE OF AIT TABLET
  Other Names: ITULATEK
  Arms: Birch allergy
Drug: GRASS 2800 BAU — DAILY DOSE OF AIT TABLET
  Other Names: GRASTEK
  Arms: Grass allergy
Drug: RAGWEED 12 AMB A 1-U — DAILY DOSE OF AIT TABLET
  Other Names: RAGWITEK
  Arms: ragweed allergy
Drug: HDM 12 SQ-HDM — DAILY DOSE OF AIT TABLET
  Other Names: ACARIZAX
  Arms: House dust mite allergy

SUMMARY:
To evaluate the tolerability of the vestibular administration route of birch pollen, grass pollen, ragweed pollen, and house dust mite (HDM) AIT tablets compared with the sublingual route in adult subjects with allergic rhinitis/conjunctivitis (AR/C)

DETAILED DESCRIPTION:
This is a single-center randomised controlled pilot trial conducted in Canada. Subjects will be randomised (1:1) to receive vestibular or sublingual birch pollen, grass pollen, ragweed pollen, or HDM AIT in tablet form for 28±4 days, followed by 28±4 days of sublingual administration only. The ratio will be ~ 1:1:1:1 for tree-, grass-, ragweed-pollen and HDM AIT tablet treatments, with a minimum of 30 patients in each allergen group for a total of approximately 200 randomised subjects.

Adults (18-65 years of age) who demonstrate birch, grass, ragweed, or HDM allergen skin prick test (SPT) positivity and with a history of birch pollen-, grass pollen-, ragweed pollen-, or HDM allergen-induced AR/C, with or without asthma are eligible for the trial.

Data for the primary endpoint of severity of treatment-related AEs will be collected during the first 28±4 days of treatment. The trial consists of 3 trial periods: a screening period (up to 12 weeks), a randomised two-arm treatment period of 28±4 days, and a single-arm sublingual treatment follow-up period of 28±4 days.

Screening period: Subjects will be evaluated based on eligibility criteria at visit 1 (V1).

Treatment period: the randomisation visit will be performed (V2) and eligible subjects randomised in a 1:1 ratio to vestibular or sublingual AIT tablet with the appropriate allergen for their allergen sensitization. At day 28±4, a visit will be conducted (V3) for all subjects previously receiving vestibular AIT to be switched to sublingual AIT with the appropriate allergen for their allergen sensitization. Subjects previously receiving sublingual AIT will remain on their previous treatment. All subjects will discontinue treatment after 56±8 days on treatment (V4). Subjects who would like to continue the sublingual immunotherapy tablets will be permitted to do so based on physician judgment and own expense but will no longer be part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial related procedures are performed

  * Male or female of any race/ethnicity aged 18-65 years at the time of signing the informed consent
  * A clinically relevant history of birch pollen-, grass pollen-, ragweed pollen-, or HDM allergen-induced AR/C with or without asthma requiring treatment during the respective allergen season for birch pollen, grass pollen, or ragweed pollen, or perennial AR/C for HDM.
  * Positive SPT (5 mm wheal size or greater) to birch pollen, timothy grass pollen, ragweed pollen, or Dermatophagoides pteronyssinus/farinae within the previous 12 months
  * A device with daily access to the internet

Exclusion Criteria:

* • Previous SLIT-tablet treatment

  * Subcutaneous AIT treatment for the sensitized allergen within less than 5 years of screening
  * Severe acute or chronic oral inflammation. Subjects with acute oral inflammation may be randomised when the condition has been resolved
  * A history or diagnosis of eosinophilic oesophagitis
  * A relevant history of systemic allergic reaction e.g. anaphylaxis with cardiorespiratory symptoms, generalised urticaria or severe facial angioedema that in the opinion of the investigator may constitute an increased safety concern
  * Unstable, severe asthma (FEV1 <70% of predicted value after adequate pharmacologic treatment) at randomisation
  * Currently taking beta-blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Tolerability (severity and number of adverse events AEs) | 28 days
  To evaluate the tolerability of the vestibular administration route

CONTACTS AND LOCATIONS:
Overall Officials: Remi Gagnon, MD, Principal Investigator — Clinique Spécialisée en Allergies de la Capitale
Locations (1):
- Clinique specialisee en allergie de la capitale, Québec, Canada